CLINICAL TRIAL: NCT00569842
Title: Investigation of the Cylex® ImmuKnow® Assay
Status: Completed | Type: Observational
Sponsor: Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Other Study IDs: 0710-11/ IUCRO-0207
Record Dates: First submitted 2007-12-05; First posted 2007-12-07 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Leukemia; Non-Hodgkin's Lymphoma; Chronic Lymphocytic Leukemia; Hodgkin's Disease; Multiple Myeloma; Myelodysplastic Syndromes; Myeloproliferative Disorders; Aplastic Anemia; Chronic Myelogenous Leukemia
MeSH Terms: conditions — Leukemia; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Hodgkin Disease; Multiple Myeloma; Myelodysplastic Syndromes; Myeloproliferative Disorders; Anemia, Aplastic; Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — None to be retained.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- observational

SUMMARY:
Currently, there is no accurate way of predicting the occurrence of Graft vs Host Disease (GvHD) or infection. The purpose of this study is to analyze blood with the ImmuKnow® Assay to see if doctors can detect which patients are at risk for GvHD and for getting an infection before they occur.

ELIGIBILITY:
Inclusion Criteria:

Patients who are undergoing allogeneic HSCT using a myeloablative preparative regimen for any of the following disorders are eligible:

1. Acute leukemia
2. Non-Hodgkin's Lymphoma
3. Chronic lymphocytic leukemia
4. Hodgkin's disease
5. Multiple myeloma
6. Myelodysplastic Syndromes
7. Myeloproliferative Disorders
8. Aplastic Anemia
9. Chronic myelogenous leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are undergoing allogeneic HSCT using a myeloablative preparative regimen for any of the following disorders are eligible:
  1. Acute leukemia
  2. Non-Hodgkin's Lymphoma
  3. Chronic lymphocytic leukemia
  4. Hodgkin's disease
  5. Multiple myeloma
  6. Myelodysplastic Syndromes
  7. Myeloproliferative Disorders
  8. Aplastic Anemia
  9. Chronic myelogenous leukemia
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2007-11; Primary Completion 2010-02 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Farag, MD, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana Universtiy Simon Cancer Center, Indianapolis, Indiana, United States